CLINICAL TRIAL: NCT00318851
Title: Treatment of Carotid Stenosis With Carotid Stenting and Neurologic Protection With Pre-Procedure and Follow-Up With MRI DIffusion Imaging and Neuropsychological Testing
Brief Title: Carotid Artery Stenting With Protection Registry
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Rodney D. Raabe, MD, Providence Sacred Heart Medical Center & Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI473
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2006-03

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid Artery stenting; Stroke
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carotid Artery Stenting (Experimental)
  Interventions: Device: Carotid Stent with Distal Protection Device

INTERVENTIONS:
Device: Carotid Stent with Distal Protection Device — Carotid Stent Placement with Distal Protection
  Other Names: Carotid Artery Stenting; Neurocognitive evaluation in Carotid Artery Stenting

SUMMARY:
The purpose of this study is to evaluate ischemic events and neuropsychological changes after carotid artery angioplasty and stenting with a neuroprotection device.

DETAILED DESCRIPTION:
Stroke is the third most common cause of death in North America with approximately 750,000 new strokes reported annually, of which 150,000 are fatal. Approximately 75% of strokes occur in the distribution of the carotid arteries. Among those, a thrombotic etiology (carotid occlusive disease) is one of the most common causes. Recently published studies have shown that patients who underwent carotid stenting in combination with a cerebral protection device had better overall outcomes as related to stroke, death and MI as opposed to carotid endarterectomy. What is not known is whether protection devices which allow some particles (100 micron particle size or less) to pass through the filter or particles that embolize during placement or removal of the protection device, will have any delayed abnormal outcomes as determined by neuropsychological testing.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 90
* Symptomatic as evidenced by transient ischemic attack or non-disabling stroke in the hemisphere supplied by the target vessel within 180 days of procedure. Must have anatomic stenosis greater than 70% by ultrasound or angiography performed in previous 30 days
* Asymptomatic patients with a stenosis greater than 80% by ultrasound or angiography performed in previous 30 days
* Patient has no childbearing potential or has negative pregnancy tests within one week prior to procedure.
* Patient and patient's physician agree to have the patient return for all the required clinical contacts following study enrollment
* Patient signs informed consent
* Patient has been excluded from other multi-institutional trials

Exclusion Criteria:

* Patient has evolving stroke or intracranial hemorrhage
* Allergy to trial required medications
* Active bleeding diathesis or coagulopathy, or will refuse blood transfusions
* History of major ipsilateral stroke with sufficient atrophy to increase risk of procedure associated bleed
* Severe dementia
* Previous intracranial hemorrhage or brain surgery within the past twelve months
* Patient has any condition that precludes angiography or would make a percutaneous procedure unsafe
* Patient or family inability to understand or cooperate with study procedures
* Recent GI or remote bleed that would interfere with anti-plate therapy
* Severe vessel tortuosity or calcification that would preclude introduction of guiding catheter, guiding sheath, or stent placement
* Extensive diffuse atherosclerotic disease involving the arch or common carotid that would preclude safe introduction of catheters and sheaths for endovascular therapy
* Intraluminal filling defect
* Intracranial aneurysm greater than 6 mm, AVM, or other intracranial vascular abnormality that would preclude safe intravascular intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Number of new diffusion weighted abnormalities post-procedure | 24 hours post stent placement

SECONDARY OUTCOMES:
Neuropsychological stability or deterioration | 3 months post procedure
Neuropsychological stability or deterioration | 6 months post procedure
Neuropsychological stability or deterioration | 12 months post procedure
Acute versus delayed neuropsychological changes | 1-7 days post procedure
Acute versus delayed neuropsychological changes | 3 months post procedure
Acute versus delayed neuropsychological changes | 6 months post procedure
Acute versus delayed neuropsychological changes | 12 months post procedure
Stroke and death | 1 month
Stroke and death | 6 months
Stroke and death | 12 months
NIH stroke scale changes | 24 hours post procedure
NIH stroke scale changes | 1 month post procedure
NIH stroke scale changes | 6 months post procedure
NIH stroke scale changes | 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rodney D. Raabe, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Sacred Heart Medical Center, Spokane, Washington, United States